CLINICAL TRIAL: NCT03103191
Title: Diagnostic Value of KL-6 in Interstitial Lung Diseases
Brief Title: Diagnostic Value of KL-6 in ILD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-KLS-2016-39
Record Dates: First submitted 2017-03-23; First posted 2017-04-06 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: * 50 subjects with fibrosing interstitial lung disease.
  * 50 subjects with pulmonary fibrosis secondary to collagen diseases.
  Interventions: Diagnostic Test: KL-6 levels
- Control: * 75 subjects without pulmonary fibrosis but with other common respiratory diseases like asthma, COPD or bronchiectasis.
  * 75 subjects with collagen disease without pulmonary fibrosis.
  Interventions: Diagnostic Test: KL-6 levels

INTERVENTIONS:
Diagnostic Test: KL-6 levels — Measure of KL-6 in serum

SUMMARY:
KL-6 may be a useful biomarker in patients with interstitial lung disease, but there is limited information in non-Asian populations. Therefore, it is necessary to carry out studies in other populations to confirm the diagnostic values of the biomarker and its prognostic implication.

Hypothesis KL-6 may be a useful biomarker in the management of interstitial lung diseases. But it is necessary to know more about its utility in the European population.

Study Objectives:

* To determine the concentration of KL-6 in serum of patients with pulmonary fibrosis at the time of diagnosis compared to patients without pulmonary fibrosis
* Diagnostic yield of KL-6 in patients with pulmonary fibrosis.
* Correlation of KL-6 values with functional and radiological parameters of disease severity at diagnosis.
* Correlation of serum KL-6 values with the evolution of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects older than 18 years.
2. Chronic respiratory diseases )including Fibrotic interstitial lung disease, asthma or COPD) related or not to a connective tissue disease.
3. Acceptance of the patient to participate in the study by signing the informed consent after having discussed with the researchers the objectives, risks and potential benefits.

Exclusion Criteria:

1. Absence of informed consent
2. Psychiatric disorder or limitation of collaboration (including language, socio-cultural problem, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects over 18 years of age attending the outpatient clinic at Hospital de la Santa Creu i Sant Pau.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-06; Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Serum KL-6 levels in patients with pulmonary fibrosis at the time of diagnosis. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain